CLINICAL TRIAL: NCT02881749
Title: Phase II Study of Low Dose Total Skin Electron Beam Treatment (TSEBT) Followed by Maintenance Valchlor for Patients With Mycosis Fungoides
Brief Title: Low Dose Total Skin Electron Beam Treatment (TSEBT) Followed by Maintenance Valchlor for Patients With Mycosis Fungoides
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #16C.514
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Mycosis Fungoides; Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — Amines

ARMS (1):
- TSEBT & mechlorethamine gel 0.016% (Experimental): All subjects enrolled in the study will receive two weeks of low dose total skin electron beam therapy (TSEBT) (12 Gy total divided into 6 fractions delivered over two weeks) followed by a weekly maintenance mechlorethamine gel 0.016% regimen for one year. The initiation of the mechlorethamine gel regimen is dependent on their disease stage downgrading to IA and IB following low dose TSEBT.
  Interventions: Radiation: Total skin electron beam therapy (TSEBT); Drug: mechlorethamine gel 0.016%

INTERVENTIONS:
Radiation: Total skin electron beam therapy (TSEBT) — TSEBT will be given in 6 fractions at 2 Gy per fraction every Monday, Wednesday, and Friday over the course of 2 weeks (total TSEBT dosage is 12 Gy). Supplements up to 8 Gy will routinely be applied to the perineum and soles as well as any other "shadowed" sites involved by disease, such as the inframammary regions, scalp, etc. Discrete tumors may receive additional "boost" up to 8 Gy.
Drug: mechlorethamine gel 0.016% — The maintenance period for this study includes one year of weekly mechlorethamine gel 0.016%. This period will not begin until the observation period (30 days) has been completed. During the first week of the maintenance period, patients will apply mechlorethamine gel to the entire body surface daily. After the first week, patients will apply mechlorethamine gel to entire body surface one time per week for the rest of the maintenance period.
  Other Names: Valchlor

SUMMARY:
The clinical efficacy of mechlorethamine gel (Valchlor) as a maintenance therapy after low dose total skin electron beam therapy (TSEBT) for the treatment mycosis fungoides cutaneous T-cell lymphoma will be evaluated in this study. Subjects will be treated with low dose TSEBT (12 Gy total) over a period of two weeks. After a 30 day observation period and confirmation that their disease stage has been downgraded to IA or IB, subjects will use Valchlor as a maintenance therapy over the course of one year. The efficacy of Valchlor as a maintenance drug will be followed clinically through Modified Severity Weight Assessment Tool (mSWAT) and percent body surface area measurements (%BSA). Furthermore, subjects will be followed histopathologically through skin biopsies performed at the screening visit, immediately after observation period, one month after the start of the maintenance period, and twelve months after the start of the maintenance period (4 biopsies total).

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or Female
* ≥ 18 years of age
* Documentation of diagnosis as evidenced by one or more clinical features consistent with Mycosis Fungoides cutaneous T-Cell lymphoma
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with requirements of the study
* Skin biopsy specimen of representative lesion obtained at screening of study and deemed diagnostic of Mycosis Fungoides by principal investigator
* Eligible, in the opinion of the investigator, for low dose TSEBT over the course of two weeks.
* Availability of subject to be observed for up to 18 months post-screening evaluation.
* Life Expectancy greater than 6 months

Exclusion Criteria:

* Pregnant or breast-feeding females
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data
* Patients diagnosed with Sezary Syndrome. Sezary Syndrome is equivalent to mycosis fungoides that develops to Stage IVA/B with B2 (high blood tumor burden) involvement, and as such requires a more aggressive treatment regimen than Valchlor or TSEBT.
* Patients who do not have their disease downgrade to stage IA or IB 30 days following low dose TSEBT.
* Underlying medical condition including unstable cardiac disease, or other serious illness that would impair the ability of the patient to undergo treatment
* Minimum 3 weeks since prior systematic treatment or phototherapy
* Decisionally-impaired individuals, prisoners, and vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Time to progression | One year
  To assess the time to progression of patients treated with total skin electron beam therapy (TSEBT) followed by the year-long maintenance Valchlor regimen.

SECONDARY OUTCOMES:
Response rate (CR and PR) | One year
  To assess the response rate (CR and PR) of patients treated with total skin electron beam therapy (TSEBT) followed by the year-long maintenance Valchlor regimen. . CR and PR are defined as the standard oncology criteria for complete response (100% reduction from the baseline score) and partial response (50% to <100% reduction from the baseline score).